CLINICAL TRIAL: NCT00945412
Title: Topical Microporous Polysaccharide Hemospheres Versus Electrocautery for Control of Pediatric Post-Tonsillectomy Bleeding
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: PI moving to another institution
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Michael J. Cunningham, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09-04-031
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2010-12

CONDITIONS: Obstructive Sleep Disorder; Obstructive Sleep Apnea; Tonsillar Hypertrophy
Keywords: microdebrider tonsillotomy; Post-tonsillectomy hemorrhage
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Electrocoagulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Micropolysaccharide Hemospheres (MPH) (Experimental)
  Interventions: Device: Micropolysaccharide Hemospheres (Arista)
- Electrocautery (Active Comparator)
  Interventions: Device: Electrocautery (Monopolar suction cautery)

INTERVENTIONS:
Device: Micropolysaccharide Hemospheres (Arista) — MPH is applied as an aerosolized powder which is applied to the bleeding fossa, immediately after suctioning the freshly completed tonsillotomy site to expose the tonsil bed. A separate aerosolizer is used for each patient in order to maximize uniformity per standard dose applied. Each initial dose remains in situ for up to 60 seconds in an attempt to achieve complete hemostasis with a single dose. (Prior data from MPH use has shown that 30-60 seconds is the time typically required for hemostasis for diffuse, non-arterial bleeds.) If there is persistent bleeding after this timeframe, then the bed is irrigated and suctioned and a second equivalent dose is applied.
  No pressure pack and no oxymetazoline or other topical vasoconstrictor is applied in either group during these initial hemostatic steps, since they are potential confounders of hemostatic effect.
  Other Names: Arista
  Arms: Micropolysaccharide Hemospheres (MPH)
Device: Electrocautery (Monopolar suction cautery) — Monopolar suction electrocautery is used at 20 Watts. Cautery is applied with a light surface touch until bleeding has stopped. In addition, any prominent visible vessels are cauterized.
  Other Names: Monopolar suction cautery
  Arms: Electrocautery

SUMMARY:
The ultimate goal of this work is to establish a method for control bleeding after tonsillectomy in awake children. Treatment of post-tonsillectomy bleeding in children typically requires general anesthesia with currently used electrocautery techniques. Micropolysaccharide hemosphere technology is a unique absorbable agent that helps clot form. These hemospheres consist of 100% purified plant starch that enhances natural clotting by concentrating blood solids such as platelets, red blood cells, and blood proteins on the particle surfaces to form a gelled matrix. This device provides painless, non-irritating control of bleeding, and has been used effectively for control of nosebleeds in awake adult patients. This device, however, has not been tested in the tonsillar fossae in children; thus, this study is performed to determine if at least 50% of children with bleeding tonsillar fossae can be spared rescue treatment with electrocautery.

ELIGIBILITY:
Inclusion Criteria:

Eligibility is contingent on the presence of following characteristics:

1. Children and adolescents age 5-18 years old. The lower age range is chosen in order to spare younger, smaller children who have less circulating volume to decrease any potential unwarranted risks of increased bleeding. The upper age range is chosen because our ultimate focus is to determine whether this therapy can help the pediatric population prevent the need for electrocautery under anesthesia for tonsil-related bleeding.
2. Obstructive sleep disorder symptomatology requiring surgical intervention. The presence of obstructive sleep disorder is determined according to the practice of the otolaryngologist investigator, and includes at least two of the following: medical history, physical exam findings, nasopharyngoscopy, lateral x-ray, sleep videotape, or polysomnography. In addition, the mean survey score on the OSD-6 (which is an instrument validated in children with obstructive sleep disorder (See Figure 2)) is at least 3, which corresponds to a moderate degree of symptoms (0 no symptoms, 6 symptoms could not be worse).
3. Tonsillar or adenotonsillar hypertrophy. Tonsillar hypertrophy is defined as at least 3+ tonsillar hypertrophy on a scale of 1+ to 4+, with the following definition of grades of obstruction determined by visual inspection: 1+ 0-25%, 2+ 26-50%, 3+ 51-75%, 4+ 76-100%.
4. Bilateral microdebrider tonsillotomy. This method of surgery is chosen because it (1) is a standard technique utilized by the surgeons involved in this study as treatment of obstructive tonsillar hypertrophy and (2) results in a relatively uniform, reproducible bleeding surface that requires hemostasis following tonsil removal.

Exclusion Criteria:

Eligibility is contingent on the absence of following characteristics:

1. Personal or family history of bleeding diathesis or easy bruising. The introduction of this confounder should be avoided, given that the primary outcome is adequacy of hemostasis. Given that preoperative laboratory evaluation in the setting of no suggestive history has been shown to have low predictive values for successful perioperative hemostasis, enrolled subjects receive no preoperative laboratory screening.
2. Intake of non-steroidal anti-inflammatory drugs within 14 days prior to surgery. Although there are several trials that suggest that postoperative administration of these drugs may have no impact on hemorrhage, the topic remains controversial due to the large numbers of subjects required to achieve adequate power in such studies. Thus, the introduction of this potential confounder is avoided, given that the primary outcome is adequacy of hemostasis.
3. Liver dysfunction. This disease state may also confound evaluation of hemostasis.
4. Cardiac, renal, or blood pressure disorder. These states may make children less tolerant of hemorrhage, and so they are excluded in order to minimize risk.
5. Chronic inflammation states, such as recurrent pharyngitis, may result in an increased propensity toward bleeding, and thus subjects with this potential confounder are excluded. Children with 3 or more acute pharyngitis episodes within the past year are excluded. A pharyngitis episode is defined as documentation by physician of the episode and >1 of the following: oral >38.3 degrees C, lymphadenopathy >2cm or tender lymphadenopathy, tonsil/pharyngeal exudates, group A beta hemolytic streptococcus positive, or antibiotic administration for proved/suspected streptococcal infection.
6. Implant contraindications to the use of monopolar electrocautery. Metal implants would preclude safe randomization to the electrocautery treatment arm. There are no suspected or known contraindications to application of MPH at the tonsillar fossae.
7. Allergic or adverse reactions to requisite perioperative medications. The current protocol calls for the use of an antibiotic and narcotic pain medication in all subjects, with one second-line agent as a planned alternative. Thus, inability to tolerate both penicillin and macrolide antibiotics, or both oxycodone and codeine narcotics, precludes entry into the trial.
8. Children whose caregivers cannot commit to the 2 week follow up schedule. This schedule includes daily calls to evaluate bleeding and pain control.
9. Cognitive inability to report bleeding, adverse events, or pain control. Thus, children with mental retardation, communication disorders, developmental delay, and chronic pain states are also excluded.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2011-06 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measure: Adequacy of intraoperative hemostasis, as evaluated by the following metrics: 1. Requirement for rescue hemostasis. 2. Time to complete hemostasis. | 0-14 days postoperatively

SECONDARY OUTCOMES:
The main secondary outcome measure is the number of patients with adverse events. These adverse events are expected to occur in the following forms: postoperative primary hemorrhage, postoperative secondary hemorrhage, and severe postoperative pain. | 0-14 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Cunningham, MD, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States